CLINICAL TRIAL: NCT00390312
Title: Randomized, Double-Blind, Placebo Controlled, Dose Ranging, Single Dose Comparison of Analgesic Efficacy and Safety of Intranasal Morphine, Immediate Release Oral Morphine, Intravenous Morphine and Placebo in Postsurgical Dental Pain
Brief Title: Efficacy and Safety of Intranasal Morphine for Pain After Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Amy Cohen/Director, Clinical Operations, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR-001
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Post-Operative Pain; Third Molar Extraction
Keywords: Post operative pain; Third molar extraction; Dental surgery; Morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 4 (Active Comparator): Intravenous morphine
  Interventions: Drug: Intravenous morphine
- 1 (Experimental): Intranasal morphine 7.5 mg
  Interventions: Drug: Intranasal morphine 7.5 mg
- 2 (Experimental): Intranasal morphine 15 mg
  Interventions: Drug: Intranasal Morphine 15 mg
- 3 (Active Comparator): Oral morphine 60 mg
  Interventions: Drug: Immediate Release Oral Morphine 60 mg
- 5 (Placebo Comparator): Intranasal placebo
  Interventions: Drug: Intranasal Placebo
- 6 (Placebo Comparator): Oral placebo
  Interventions: Drug: Oral placebo
- 7 (Placebo Comparator): Intravenous placebo
  Interventions: Drug: Intravenous placebo

INTERVENTIONS:
Drug: Intranasal Placebo — Intranasal placebo
  Arms: 5
Drug: Intranasal Morphine 15 mg — Intranasal Morphine 15 mg
  Arms: 2
Drug: Immediate Release Oral Morphine 60 mg — Immediate Release Oral Morphine 60 mg
  Arms: 3
Drug: Intravenous morphine — Intravenous morphine 7.5 mg
  Arms: 4
Drug: Intranasal morphine 7.5 mg — Intranasal morphine 7.5 mg
  Arms: 1
Drug: Oral placebo — Oral placebo
  Arms: 6
Drug: Intravenous placebo — Intravenous placebo
  Arms: 7

SUMMARY:
This study involves approximately 200 patients designed to evaluate the efficacy and safety of intranasal (IN) morphine 7.5 mg and 15 mg, intravenous morphine (IV) 7.5 mg, immediate release oral (PO) morphine 60 mg or placebo in patients with acute postsurgical pain following third molar extraction.

DETAILED DESCRIPTION:
Diagnosis and Main Criteria for Inclusion: Dental outpatients undergoing the removal of 3 or more third molars (2 of which were required to be mandibular and both must be bony impacted third molars).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-40 years of age
* Surgical extraction of at least three or more third molars (two must be mandibular and both must be bony impacted third molars)
* Moderate or severe pain within 6 hours of completion of surgery

Exclusion Criteria:

* Other oral surgical procedures during the same session except the removal of supernumerary third molars
* Evidence of nasal congestion, nasal polyps, mucosal lesions of the nostrils, postnasal drip of any etiology or any clinically significant nasal pathology that may affect the absorption of study medication or the assessment of safety
* Chronic respiratory insufficiency such that treatment with an opioid analgesic is contraindicated
* Allergy to shellfish

Additional Inclusion/Exclusion Criteria May Apply

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2001-09; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Total pain relief (TOTPAR) at the 0-2 hour time interval calculated as the time-weighted sum of the Pain Relief (PR) scores for the time interval 0-2 hours | 2 hours

SECONDARY OUTCOMES:
Other measures of pain relief | Several time points

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Christensen, DDS, Principal Investigator — Jean Brown Associates, Inc.